CLINICAL TRIAL: NCT05767060
Title: A Multi-center, Open Phase Ia/Ib Clinical Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Preliminary Clinical Efficacy of BAT7104 Injection in Patients With Advanced Malignant Tumors.
Brief Title: BAT7104 Injection in Patients With Advanced Malignant Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-7104-001-CR
Record Dates: First submitted 2023-02-10; First posted 2023-03-14 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- BAT7104 Injection 0.1 mg/kg (Experimental): frequency: Q2W
  Interventions: Drug: BAT7104 injection
- BAT7104 Injection 0.3 mg/kg (Experimental): frequency: Q2W
  Interventions: Drug: BAT7104 injection
- BAT7104 Injection 1 mg/kg (Experimental): frequency: Q2W
  Interventions: Drug: BAT7104 injection
- BAT7104 Injection 3 mg/kg (Experimental): frequency: Q2W
  Interventions: Drug: BAT7104 injection
- BAT7104 Injection 10 mg/kg (Experimental): frequency: Q2W
  Interventions: Drug: BAT7104 injection
- BAT7104 Injection 20 mg/kg (Experimental): frequency: Q2W
  Interventions: Drug: BAT7104 injection
- BAT7104 Injection 40 mg/kg (Experimental): frequency: Q2W
  Interventions: Drug: BAT7104 injection

INTERVENTIONS:
Drug: BAT7104 injection — According to the protocol, each dose group is given intravenous infusion at the rate of mg/kg, and the recommended infusion time is ≥ 60 minutes. Once every two weeks (Q2W), on the first day of each cycle.
  Other Names: Recombinant anti-PD-L1/CD47 bispecific antibody injection

SUMMARY:
A multi-center, open phase Ia/Ib clinical study to evaluate the safety, tolerance, pharmacokinetics and preliminary clinical efficacy of BAT7104 injection in patients with advanced malignant tumors.

DETAILED DESCRIPTION:
This is a multi-center, open, dose-increased and dose-expanded phase I clinical study. About 18-42 patients will be recruited from research centers in China. In the stage of dose increase, the safety, tolerance, pharmacokinetics and preliminary clinical efficacy of BAT7104 injection in patients with advanced malignant tumors were investigated by using accelerated titration and "3+3" dose increase design. During the dose increase test, the appropriate dose was selected according to the previous study data of the extended study.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old and ≤ 80 years old, gender: male or female;
2. The investigator evaluated the expected survival period to be at least 3 months;
3. The requirement of the ECOG physical fitness score is 0 or 1;
4. Patients with advanced malignant tumors who have failed to receive standard treatment, have no standard treatment, do not tolerate standard treatment or refuse to accept standard treatment confirmed by cytology or pathology;
5. There must be an evaluable tumor focus in the dose increasing stage, and at least one measurable tumor focus in the dose expanding stage (solid tumors refer to RECIST 1.1 standard, lymphoma refer to Lugano 2014 evaluation standard);
6. It has sufficient organ and bone marrow reserve function, which is defined as follows:

   System laboratory reference value:

   Blood routine (no blood transfusion, no use of hematopoietic stimulating factor and no use of drugs to correct blood cell count within 14 days before the first administration):

   Absolute neutrophil count ≥ 1.5 x 109/L;Platelet count ≥ 90 x109/L;Hemoglobin ≥ 90g/L;

   Coagulation function:

   International standardized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5xULN (without anticoagulant treatment), those who receive oral anticoagulant treatment and whose INR is 2~3 can be included.

   Liver function:

   Total bilirubin (TBIL) ≤ 1.5xULN;Hepatocellular carcinoma, Gilbert's syndrome, liver metastasis ≤ 2xULN;Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5xULN;Hepatocellular carcinoma, liver metastasis ≤ 5xULN renal function Serum creatinine or Serum creatinine clearance ≤ 1.5xULN or>50ml/min (using Cockcroft-Gault formula, see appendix)
7. Agree to provide archived pathological tissue or fresh biopsy tumor tissue for the detection of PD-L1, CD47 expression level or receptor occupancy and other pharmacodynamic indicators (not as a necessary inclusion standard); Female patients with fertility must have negative serum pregnancy test within 7 days before the first administration and are willing to take effective birth control/contraception methods to prevent pregnancy during the study period until 6 months after the last administration of the study. Male patients must agree to take effective contraceptive methods during the study period and within 6 months after the last administration of the study; Postmenopausal women must have amenorrhea for at least 12 months before they are considered infertile.

Exclusion Criteria:

1. Have received any anti-CD47 antibody and SIRP within 4 weeks before the first administration α Antibodies or CD47/SIRP α Recombinant protein therapy;
2. He has received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy and other anti-tumor treatment within 4 weeks before the first use of the study drug, with the exception of the following: ① nitrosourea or mitomycin C within 6 weeks before the first use of the study drug; ② Oral fluorouracil and small-molecule targeted drugs are 2 weeks before the first use of the study drug or within 5 half-lives of the drug (whichever is longer); ③ The systematic treatment of traditional Chinese medicine/proprietary Chinese medicine with clear anti-tumor effect and drugs with immunomodulatory effect (including but not limited to thymosin, interferon, interleukin, etc.) is within 2 weeks before the first use of the study drug;
3. Those who are participating in or have participated in the experimental drug or medical device intervention clinical research within 4 weeks before the first administration of this study cannot be included; In the survival follow-up stage of the intervention study, if the time between the first administration and the end of the previous study (the last administration) meets the above exclusion criteria, it can be included;
4. Inoculated or planned to receive live/attenuated vaccine and mRNA vaccine within 4 weeks before screening;
5. Pregnant or lactating women;
6. AEs caused by previous anti-tumor therapy are still higher than grade 1 (based on CTCAE v5.0) before the first administration of the study drug (except for AEs such as hair loss and fatigue that cannot be restored to ≤ grade 1 and will remain stable for a long time according to the judgment of the researcher based on clinical actual conditions, except for grade 2 peripheral neurotoxicity, and hypothyroidism stabilized by hormone replacement therapy);
7. Those who have had ≥ 3 levels of irAE in the past or have terminated immunotherapy due to any level of irAE;
8. Primary central nervous system tumor, central nervous system metastasis with related symptoms, meningeal metastasis or previous history of epilepsy should be excluded. Patients with asymptomatic or asymptomatic central nervous system metastasis who have been clinically controlled but have been judged stable by the researcher can be included, but the following conditions must be met at the same time: a The disease was stable ≥ 4 weeks before the first administration; B. No evidence of central nervous system disease progression was found in MRI enhancement of the head within 4 weeks before the first administration; C. The anticonvulsant drugs have been stopped at least 2 weeks before the first administration, and the dosage of prednisone is ≤ 10mg/day or equivalent dose of hormone;
9. Patients who have undergone major organ surgery (excluding puncture biopsy) or had significant trauma within 4 weeks before the first use of the study drug, or who need to undergo elective surgery during the trial period;
10. Have a history of tissue or organ transplantation;
11. Patients with severe infection within 4 weeks before the first medication, including but not limited to infection complications, bacteremia, severe pneumonia, etc. requiring hospitalization; Patients with active infection before the first administration were excluded;
12. Known history of human immunodeficiency virus (HIV) infection;
13. Active hepatitis B, untreated chronic hepatitis B or treated but uncontrolled chronic hepatitis B (HBV DNA>200 IU/mL or>103 copies/ml);
14. Active HCV infected patients (HCV antibody positive and HCV-RNA level higher than the lower limit of detection);
15. Untreated or under treatment tuberculosis patients, including but not limited to tuberculosis; Those who have received standard anti-tuberculosis treatment and have been confirmed as cured by researchers can be included;
16. Known to have a history of severe allergy, or known to have had ≥ grade 3 allergic reaction to macromolecular protein preparation/monoclonal antibody, and any component of test drug;
17. Patients with active, or had a history of autoimmune diseases that may recur (excluding vitiligo, autoimmune thyroid diseases that can be treated with hormone replacement therapy, and type 1 diabetes patients);
18. Have received systemic glucocorticoid (prednisone>10mg/day or equivalent dose of the same drug) or other immunosuppressive treatment within 14 days before the first use of the study drug, except for the following cases: ① use of local, ocular, intraarticular, intranasal and inhaled glucocorticoid treatment, ② short-term use of glucocorticoid for preventive treatment (such as prevention of contrast agent allergy);
19. Patients who have a history of non-infectious pneumonia requiring glucocorticoid treatment or who currently have interstitial lung disease within 1 year before the first administration;
20. There is a history of serious cardio-cerebrovascular disease, including but not limited to: ① heart failure or left ventricular ejection fraction (LVEF)<50% with NYHA grade II or above; ② There are serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, Ⅱ - Ⅲ degree atrioventricular block, etc.; ③ Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular and cerebrovascular events of grade 3 or above occurred within 6 months before the first administration; ④ Hypertension that cannot be controlled clinically (this protocol is defined as that although antihypertensive treatment is adopted, the systolic blood pressure is more than 150 mmHg and/or diastolic blood pressure is more than 100 mmHg after treatment, and has clinical significance after evaluation by the researcher);
21. Those with the following risk of thrombosis or bleeding:

    A. Myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack occurred within 6 months before the first administration; B. There is a history of deep venous thrombosis, pulmonary embolism or any other serious thromboembolism within 3 months before the first administration (implantable venous infusion port or catheter-derived thrombosis, or superficial venous thrombosis is not considered as "serious" thromboembolism); C. Any life-threatening bleeding event or grade 3 or 4 gastrointestinal/variceal bleeding event requiring blood transfusion, endoscopy or surgical treatment within 3 months before the first administration; D. Other diseases that the researcher believes have a high risk of bleeding or thrombosis in the future;
22. Patients who are known to have a history of abuse or drug abuse of psychotropic substances and are considered to affect the compliance of this study;
23. Have a history of hemolytic anemia or Evans syndrome in the past 3 months;
24. In addition to the tumors at the time of study, there are other active malignant tumors within 3 years before the first administration (not excluding locally cured tumors, such as skin basal cell carcinoma, superficial bladder cancer cancer or breast cancer in situ);
25. Patients with pleural effusion, pericardial effusion or ascites that are not controlled or need drainage;
26. Patients who are not suitable for this study according to the researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT), | A minimum of 28 days after first dose of BAT-7104
  umber of subjects who experience DLT events during 28 days. Toxicity will be graded according to CTCAE, Version 5.0.
Adverse Events (AEs) | AE needs continuous monitoring and evaluation from the first administration to 90 days after the last administration or before receiving new anti-tumor treatment.
  Incidence of treatment -related AEs as assessed by CTCAE, Version 5.0.

SECONDARY OUTCOMES:
Cmax, | up to Cycle 6, each cycle is 14 days
  Maximum observed plasma or serum concentration
Anti-drug antibodies (ADA) and neutralizing antibodies (NAb) | up to Cycle 6, each cycle is 14 days
Objective response rate (ORR) | 12 months (anticipated)
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Tmax (Time to reach maximum serum concentration) | up to Cycle 6, each cycle is 14 days
  Time to Maximum concentration
AUC0-inf after Cycle 1 administration and AUC0- λ after Cycle 6 administration | up to Cycle 6, each cycle is 14 days
Systemic Clearance (CL) | up to Cycle 6, each cycle is 14 days
  Systemic dose clearance
Vss (volume of distribution at steady state) | up to Cycle 6, each cycle is 14 days
  Amount of drug in the body divided by plasma concentration
t1/2 (terminal half-life) | up to Cycle 6, each cycle is 14 days
  Apparent terminal-phase disposition half-life.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Li Zhang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No